CLINICAL TRIAL: NCT06866821
Title: Comparison of Mulligan's Spinal Mobilization With Proprioceptive Neuromuscular Facilitation Technique on Pain, Disability and Range of Motion in Patients With Cervical Radiculopathy
Brief Title: Spinal Mobilization and PNF Comparison on Pain, Disability in Patients With Cervical Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Muhammad Azeem
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Cervical Radiculopathy
Keywords: Cervical Radiculopathy; Pain; Range of Motion; Distraction; Proprioceptive Neuromuscular Facilitation
MeSH Terms: conditions — Radiculopathy; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (SMWAM's and PNF C-R Technique) (Experimental): Experimental group received Mulligan's Spinal Mobilization with Arm Movements and Proprioceptive Neuromuscular Facilitation contract-relax technique.
  Interventions: Other: SMWAM's and PNF C-R Technique
- Control Group (PNF C-R Technique and PT Protocol) (Experimental): Control group received Proprioceptive Neuromuscular Facilitation Contract-relax Technique and Physical Therapy protocol.
  Interventions: Other: PNF C-R Technique and PT Protocol

INTERVENTIONS:
Other: SMWAM's and PNF C-R Technique — Treatment provided 3 days every week in 6 total weeks with 1 meeting per day, 3 bunches of 10 times repeat and resting period of one minute among bunches. This group received Mulligan's spinal mobilization with arm movement and proprioceptive neuromuscular facilitatin contract-relax technique. Previous to mobilization, all patients got hot pack (10 minutes) and active range of motion warm up exercises (2 sets of 10 repetitions) and did isometric neck exercise as a home plan of care.
  Mobilisation (22) was done depending on the side of involvement, the corresponding spinous process would be mobilised combined with different movements of shoulder (flexion/ abduction/ horizontal abduction/ horizontal adduction).
  Proprioceptive neuro-muscular facilitation contract relax technique performed with 3 repetitions in each cervical movement (flexion, extension, lateral flexion and rotation) (27).
  Arms: Experimental Group (SMWAM's and PNF C-R Technique)
Other: PNF C-R Technique and PT Protocol — Treatment provided 3 days every week in 6 weeks with 1 meeting per day, 5 clusters of 3 times repeat and resting period of one minute among clusters. Regime of training involved PNF (proprioceptive neuromuscular facilitation) contract-relax method along with the standard physical therapy protocol which includes passive stretching (3 sets of 10 repetitions) and isometric strengthening exercises (2 sets of 10 repetitions).
  Proprioceptive neuro-muscular facilitation contract relax technique performed with 3 repetitions in each cervical movement (flexion, extension, lateral flexion and rotation) (27).
  Arms: Control Group (PNF C-R Technique and PT Protocol)

SUMMARY:
As in this modern era of digitalization; mobile phones, touch pads and computers devices use is increasing, neck pain that radiates into upper limb is also becoming common due to such devices long term use in bad postures or positions for more workload. The resulted findings could significantly contribute to the refinement of rehabilitation interventions, offering a more holistic and tailored approach for addressing cervical radiculopathy sensory and motor symptoms, ultimately improving individuals daily living activities and life quality. It will be helpful for physiotherapists to find evidence about comparison of mulligan's spinal mobilization along with arm movement with proprioceptive neuromuscular facilitation technique on pain, disability and range of motion in patients with cervical radiculopathy. It will be beneficial for patients also to improve pain, activities of daily living and working tasks in a comfortable position.

DETAILED DESCRIPTION:
Cervical radiculopathy is a clinical situation in which reflex, motor, and sensory alterations e.g. radicular pain, paresthesia, or numbness might be present and might be increased by neck bad postures and movements. Due to sustained forward head and neck posture and repetitive movements, cervical pain and numbness is becoming common in office, bank and online workers. The cervical radiculopathy new cases report yearly is almost 107.3 per 1 lac for men and 63.5 per 1 lac for women. It is essential to find new efficient methods of cervical radiculopathy physical therapy management.

Males and females of age 21-50 years old added in this study. Screening tests will include upper limb tension tests (ULTT), spurling (compression) test and distraction test. Subjects randomly assigned into two groups by lottery method. Experimental group (N=19) received Mulligan's spinal mobilization with arm movements (SMWAMs) and proprioceptive neuromuscular facilitation (PNF) contract-relax technique and control group (N=19) received Proprioceptive neuromuscular facilitation (PNF) contract-relax technique and standard physical therapy protocol including passive stretching exercises (3 sets of 10 repetitions) and isometric strengthening exercises (2 sets of 10 repetitions). Outcome measures included numeric pain rating scale (NPRS) for pain, neck disability index (NDI) for functional disability and goniometer for range of motion (ROM). Data analyzed by statistical package for social sciences (SPSS 26) software.

ELIGIBILITY:
Inclusion Criteria:

* Both males, females of 21 years to 50 years old
* Patients already diagnosed by orthopedicians
* Patients with positive screening (upper limb tension, spurling & distraction) tests

Exclusion Criteria:

* History of trauma, fracture and previous surgery
* Any pathological condition, spinal instability and tumor
* VBI (Vertebral-Basillar Insufficiency) and cervical instability/spondylolisthesis

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Males and Females
Enrollment: 38 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Pain by Numeric Pain Rating Scale | 6 weeks
  This was used for pain intensity assessment. Patient rested on stool or chair and ordered to score resting pain extent in between 0 and 10 range; 0 means without pain and 10 means much high pain as possible in 10cm numbers line.
Neck level of disability by Neck Disability Index | 6 weeks
  Neck disability Index was used for functional disability of neck assessment. NDI is a 10-items questionnaire that assesses the effect of neck signs and symptoms on daily living functional activities. Every item is marked from range 0 to 5, along with total score from 0 to 50 range and maximum scores means maximum disability. NDI has reliability acceptable in the self-perceptual disability assessment and an MCID (minimal clinically important difference) of 8.5 points in cervical radiculopathy patients.
Cervical Range of Motion by Goniometer | 6 weeks
  Goniometer was used for active cervical spine range of the motion (flexion, extension, rotation, side bending) assessment. Side bending, rotation measured on the symptomatic and asymptomatic both sides.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Azeem, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kamal AS, Zakaria HM, Elsamra MK, Gaballah MA, Elrewainy RM. EFFICACY OF PROPRIOCEPTIVE TRAINING PARADIGM ON CERVICAL RADICULOPATHY. Assessment. 2023;1000(2):12.
- [Background] Gashi AI, Kovačič T, Gashi F, Azemi A. The effect of proprioceptive neuromuscular facilitation technique on treating cervical radiculopathy. Journal of Physical Education and Sport. 2023;23(3):722-9.
- [Background] Taneja D, Saharan A, Ranjeeta W, Sharma M, Saharan M, Dubey S, et al. Effect of Mulligan's Smwam among Subjects with UnilateralCervical Radiculopathy. Eduzone: International Peer Reviewed/Refereed Multidisciplinary Journal. 2023;12(1):11-22.